CLINICAL TRIAL: NCT04553549
Title: Safety and Feasibility of the Infinity Guide Catheter for Neuro Interventional Procedures Using Transradial Access
Brief Title: Safety and Feasibility of the Infinity Catheter for Radial Access
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Priyank Khandelwal, MD, Assistant Professor, Rutgers, The State University of New Jersey
Other Study IDs: Pro2020000869
Record Dates: First submitted 2020-08-31; First posted 2020-09-17 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Brain Tumor; Stroke, Acute; Brain Aneurysm; Intracranial Arteriovenous Malformations; Carotid Stenosis; Cavernous Sinus Thrombosis
Keywords: neuro-embolization
MeSH Terms: conditions — Brain Neoplasms; Stroke; Intracranial Aneurysm; Intracranial Arteriovenous Malformations; Carotid Stenosis; Cavernous Sinus Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Transradial approach: The procedure will be done using standard criteria as per operator preference. All interventional cases at our institution undergo a "radial first" approach, meaning that the access site of choice is the radial artery. The investigators will measure the radial artery size to ensure that the artery is greater than 2.4 mm in order to use the Infinity catheter (8Fr).
  Interventions: Device: Transradial approach

INTERVENTIONS:
Device: Transradial approach — Patients who are undergoing endovascular intervention will be enrolled into the study. As the metrics analyzed in this study are already normally collected, this study can be considered as a secondary use of the data. The procedure will be done using standard criteria as per operator preference. All interventional cases at the study institution undergo a "radial first" approach, meaning that the access site of choice is the radial artery. The investigators will measure the radial artery size to ensure that the artery is greater than 2.4 mm in order to use the Infinity catheter (8Fr).

SUMMARY:
The main objective of this single arm study is to evaluate the safety and feasibility of the AXS Infinity LS (Stryker, Freemont, CA, USA) and AXS Infinity LS Plus (Stryker, Freemont, CA, USA) catheters during the transradial approach through a secondary use of the data collected during neurointerventional procedures. This includes evaluating the conversion rates to a transfemoral approach. A secondary aim of the study is to assess the radial artery occlusion rates post procedure.

DETAILED DESCRIPTION:
Patients who are undergoing endovascular intervention will be enrolled into the study. Consent will be obtained for the procedure and for the use of their prospectively collected clinical data. As the metrics analyzed in this study are already normally collected, this study can be considered as a secondary use of the data. The procedure will be done using standard criteria as per operator preference. All interventional cases at the study institution undergo a "radial first" approach, meaning that the access site of choice is the radial artery. The investigators will measure the radial artery size to ensure that the artery is greater than 2.4 mm in order to use the Infinity catheter (8Fr). If the artery does not meet the size criteria, only a 6Fr sheath will be used, and the data recorded during the procedure will not be utilized for analysis in this study. The preoperative and postoperative care will be the same for all the patients. No tests will be done outside of standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age group 18 years and above.
* Patients undergoing neuro-embolization using large bore catheters

Exclusion Criteria:

* Patients with Radial artery diameter less than 2.4 mm measured with Ultrasound
* Age<18
* Patients who have previous surgeries at either approach site which precludes the use of one of the approach sites
* Patients who has poor collateral circulation, Raynaud's phenomenon, radial loop, brachial or subclavian stenosis, aberrant origin of the subclavian artery
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing endovascular intervention will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of TRA Intervention | 1 month
  The size of the radial artery will be measured and the transradial approach will be used. Notation will be also be recorded if conversion to TFA is used.

SECONDARY OUTCOMES:
Assess radial artery occlusion rates post procedure | 1 month
  Reverse Barbue Test and ultrasound
Demographics | 1 month
  Patient demographics will be analyzed such as past medical history, HTN, HLD, Afib

CONTACTS AND LOCATIONS:
Overall Officials: Priyank Khandelwal, MD, Principal Investigator — Rutgers University
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be presented

REFERENCES:
- [Background] Jolly SS, Amlani S, Hamon M, Yusuf S, Mehta SR. Radial versus femoral access for coronary angiography or intervention and the impact on major bleeding and ischemic events: a systematic review and meta-analysis of randomized trials. Am Heart J. 2009 Jan;157(1):132-40. doi: 10.1016/j.ahj.2008.08.023. Epub 2008 Nov 1. PMID 19081409
- [Background] Bertrand OF, Rao SV, Pancholy S, Jolly SS, Rodes-Cabau J, Larose E, Costerousse O, Hamon M, Mann T. Transradial approach for coronary angiography and interventions: results of the first international transradial practice survey. JACC Cardiovasc Interv. 2010 Oct;3(10):1022-31. doi: 10.1016/j.jcin.2010.07.013. PMID 20965460
- [Background] Hamon M, Pristipino C, Di Mario C, Nolan J, Ludwig J, Tubaro M, Sabate M, Mauri-Ferre J, Huber K, Niemela K, Haude M, Wijns W, Dudek D, Fajadet J, Kiemeneij F; European Association of Percutaneous Cardiovascular Interventions; Working Group on Acute Cardiac Care of the European Society of Cardiology; Working Group on Thrombosis on the European Society of Cardiology. Consensus document on the radial approach in percutaneous cardiovascular interventions: position paper by the European Association of Percutaneous Cardiovascular Interventions and Working Groups on Acute Cardiac Care** and Thrombosis of the European Society of Cardiology. EuroIntervention. 2013 Mar;8(11):1242-51. doi: 10.4244/EIJV8I11A192. PMID 23354100
- [Background] Kolkailah AA, Alreshq RS, Muhammed AM, Zahran ME, Anas El-Wegoud M, Nabhan AF. Transradial versus transfemoral approach for diagnostic coronary angiography and percutaneous coronary intervention in people with coronary artery disease. Cochrane Database Syst Rev. 2018 Apr 18;4(4):CD012318. doi: 10.1002/14651858.CD012318.pub2. PMID 29665617
- [Background] Snelling BM, Sur S, Shah SS, Khandelwal P, Caplan J, Haniff R, Starke RM, Yavagal DR, Peterson EC. Transradial cerebral angiography: techniques and outcomes. J Neurointerv Surg. 2018 Sep;10(9):874-881. doi: 10.1136/neurintsurg-2017-013584. Epub 2018 Jan 8. PMID 29311120

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT04553549/SAP_000.pdf
  • Informed Consent Form (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT04553549/ICF_001.pdf